CLINICAL TRIAL: NCT01874405
Title: Effectiveness of Deferasirox Therapy on Comprehensive Management of Iron Overload in Adult and Pediatric Transfusion-dependent Patients: a Long Term Retrospective Study
Brief Title: Retrospective Evaluation of Adult and Pediatric Transfusion-dependent Patients Treated With Deferasirox Therapy
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Silverio Perrotta, MD, University of Campania Luigi Vanvitelli
Other Study IDs: DIPEDNA-2013-1
Record Dates: First submitted 2013-05-26; First posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Iron Overload
Keywords: Iron overload; thalassaemia; deferasirox; magnetic resonance; endocrine function
MeSH Terms: conditions — Iron Overload; Thalassemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Iron overload is a leading cause of morbidity and mortality in transfusion-dependent patients. Deferasirox is the most promising iron chelator agent in several clinical scenarios. The investigators propose a retrospective study (chart review) to evaluate comprehensive iron overload management in transfusion-dependent patients treated with deferasirox for up to 5-10 years in a real clinical practice setting.

ELIGIBILITY:
Inclusion Criteria:

* Transfusion- dependent patients (> 2 years);
* Ongoing deferasirox therapy during the study period;
* ≥ 2 Magnetic Resonance scans (one at baseline and at least one post baseline - as per clinical need) during study period (this criteria is not mandatory for patients undergoing only the endocrine subanalysis and participating only to the cardiac analysis);
* Available medical history including relevant clinical and laboratory data (e.g serum ferritin, liver function tests, renal function tests, endocrine parameters ) at baseline before starting deferasirox treatment

Exclusion Criteria:

* Non transfusion- dependent patients;
* Other chelation therapy than deferasirox;
* Absence of complete medical history as above specified

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric transfusion- dependent patients (male and female) with different underlying cronic anemias who received iron chelation therapy with deferasirox during the observational study period and underwent at least 2 cardiac MRI scans at the Pozzuoli site.
  All consecutive patients visited at the participating sites starting from March 2003 to October 2012 will be entered in this observational study (chart review) provided all the inclusion an no exclusion criteria are met.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2003-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
cardiac T2* in patients treated with deferasirox | at least 1 year
  change from baseline to end of study in cardiac T2*, as measured by Magnetic Resonance, in patients with iron overload (cardiac T2* <20 ms at baseline)
cardiac T2* in patients treated with deferasirox | at least 1 year
  maintenance from baseline to end of study of cardiac T2* in not iron overloaded patients (cardiac T2* >20 ms at baseline)

SECONDARY OUTCOMES:
cardiac function in patient undergoing deferasirox treatment | at least 1 year
  change in left and right ejection fraction, telediastolic and telesystolic volumes, stroke volumes, cardiac output, myocardial mass, measured by Cardiac Magnetic Resonance, from baseline to end of study
change in liver iron concentration | at least 1 year
maintenance of normal endocrine function in patients without endocrine dysfunction and improvement in disease severity in patients affected by endocrine dysfunction from baseline to end of study | at least 3 years
  Thyroid function (TSH, free triiodothyronine and free thyroxine serum free T4 levels), pancreatic cell function (basal glycemia, glycated hemoglobin level), bone mineral density (z-score) will be evaluated by the closest assessment to baseline (first deferasirox exposure) and to the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Silverio Perrotta, MD, Principal Investigator — University of Campania Luigi Vanvitelli

REFERENCES:
- [Derived] Casale M, Citarella S, Filosa A, De Michele E, Palmieri F, Ragozzino A, Amendola G, Pugliese U, Tartaglione I, Della Rocca F, Cinque P, Nobili B, Perrotta S. Endocrine function and bone disease during long-term chelation therapy with deferasirox in patients with beta-thalassemia major. Am J Hematol. 2014 Dec;89(12):1102-6. doi: 10.1002/ajh.23844. Epub 2014 Sep 26. PMID 25197009